CLINICAL TRIAL: NCT07232758
Title: Safety, Tolerability and Pharmacokinetic Studies of HRS-2183 for Injection in Healthy Chinese Subjects After Single and Multiple Administration
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-2183-102
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Chinese Healthy Adult Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A:HRS-2183 (Experimental)
  Interventions: Drug: HRS-2183
- Treatment group B:placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HRS-2183 — HRS-2183
  Arms: Treatment group A:HRS-2183
Drug: Placebo — placebo
  Arms: Treatment group B:placebo

SUMMARY:
This study mainly evaluated the safety and tolerability, as well as the pharmacokinetic characteristics, of the injectable drug HRS-2183 after single and multiple administrations in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects, aged 18 to 45 years.
2. Body weight and Body Mass Index (BMI) within a specified range (e.g., BMI 19.0-26.0 kg/m²).
3. Agreement to use highly effective contraception during the study period and for a specified duration after the last dose. No plans for pregnancy, sperm/egg donation.
4. Voluntarily provides written informed consent to participate in the study.

Exclusion Criteria:

1. History of significant allergies to any food or drug, especially to the investigational product, its components, or drugs of a similar class.
2. History or current presence of any clinically significant disease in major organ systems (e.g., cardiovascular, hepatic, renal, neurological, etc.).
3. Any clinically significant abnormalities found during screening assessments (including physical examination, vital signs, and laboratory tests).
4. Clinically significant abnormalities on 12-lead electrocardiogram (ECG) at screening.
5. Evidence of impaired renal function based on laboratory tests (e.g., eGFR, serum creatinine).
6. Positive screening for specified infectious diseases (e.g., HIV, HBV, HCV, Syphilis).
7. Use of any medication (including prescription, OTC, and herbal) within a specified period before the study.
8. Excessive consumption of certain beverages (e.g., caffeine, grapefruit juice) or inability to adhere to dietary restrictions.
9. History of major surgery within the past 3 months or planned surgery during the study period.
10. Participation in another clinical trial within the past 3 months.
11. Significant blood loss, blood donation, or transfusion within the past 3 months.
12. History of excessive alcohol consumption or unwillingness to abstain during the study.
13. History of heavy smoking or unwillingness to abstain during the study.
14. History of drug abuse or positive drug screening test.
15. Inability to tolerate venous access or history of fainting during blood draws.
16. Inability to comply with the standardized diet provided during the study.
17. Any other reason that, in the opinion of the investigator, makes the subject unsuitable for the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of any adverse events | Evaluation was performed up to the seventh day / the 16th day

SECONDARY OUTCOMES:
Tmax (Pharmacokinetic Parameters after a Single Dose) | Evaluation was performed up to the third day
Cmax(Pharmacokinetic Parameters after a Single Dose) | Evaluation was performed up to the third day
AUC0-t(Pharmacokinetic Parameters after a Single Dose) | Evaluation was performed up to the third day
AUC0-∞(Pharmacokinetic Parameters after a Single Dose) | Evaluation was performed up to the third day
t1/2(Pharmacokinetic Parameters after a Single Dose) | Evaluation was performed up to the third day
CLz(Pharmacokinetic Parameters after a Single Dose) | Evaluation was performed up to the third day
Vz(Pharmacokinetic Parameters after a Single Dose) | Evaluation was performed up to the third day
Ae0-t(Pharmacokinetic Parameters after a Single Dose) | Evaluation was performed up to the third day
Fe0-t(Pharmacokinetic Parameters after a Single Dose) | Evaluation was performed up to the third day
CLr(Pharmacokinetic Parameters after a Single Dose) | Evaluation was performed up to the third day
Tmax(Pharmacokinetic Parameters after Multiple Doses) | Evaluation was performed up to the 12th day
Cmin,ss(Pharmacokinetic Parameters after Multiple Doses) | Evaluation was performed up to the 12th day
Cmax,ss(Pharmacokinetic Parameters after Multiple Doses) | Evaluation was performed up to the 12th day
Cav(Pharmacokinetic Parameters after Multiple Doses) | Evaluation was performed up to the 12th day
AUC0-t,ss(Pharmacokinetic Parameters after Multiple Doses) | Evaluation was performed up to the 12th day
AUC0-τ,ss(Pharmacokinetic Parameters after Multiple Doses) | Evaluation was performed up to the 12th day
AUC0-∞,ss(Pharmacokinetic Parameters after Multiple Doses) | Evaluation was performed up to the 12th day
t1/2(Pharmacokinetic Parameters after Multiple Doses) | Evaluation was performed up to the 12th day
CLss(Pharmacokinetic Parameters after Multiple Doses) | Evaluation was performed up to the 12th day
Vss(Pharmacokinetic Parameters after Multiple Doses) | Evaluation was performed up to the 12th day
Rac(Pharmacokinetic Parameters after Multiple Doses) | Evaluation was performed up to the 12th day
DF(Pharmacokinetic Parameters after Multiple Doses) | Evaluation was performed up to the 12th day

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided